CLINICAL TRIAL: NCT04097847
Title: Osteoradionecrosis and PENTOCLO Protocol: Retrospective Study.
Acronym: OPEN
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: OPEN (29BRC17.0115)
Record Dates: First submitted 2019-05-14; First posted 2019-09-20 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-02

CONDITIONS: Osteoradionecrosis of Jaw
MeSH Terms: interventions — pentoxifylline-tocopherol-clodronate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pentoxifylline-Tocopherol-Clodronate — the aim of this retrospective study is to analyze from patient records the impact of the PENTOCLO protocol on maxillofacial osteoradionecrosis at Brest Hospital University, France.
  Other Names: Pentoclo

SUMMARY:
osteoradionecrosis (ORN) affects up to 30% of irradiated patients and can occur up to several decades after stopping treatment. Differents therapeutics exist but there is no consensus concerning the management of the maxillary ORN. The understanding of new pathological mechanisms opens the way to new therapeutic perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 being or having been treated by pentoclo combination for an osteoradionecrosis of the jaw

Exclusion Criteria:

* Tumoral recidivism
* Precocious stop of pentoclo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients treated at Brest hospital University for ENT cancer and who had cervicofacial radiotherapy, with maxillary and / or mandibular osteoradionecrosis treated with PENTOCLO alone or in combination with other therapies
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical evolution of the osteoradionecrosis lesion after introducing PENTOCLO protocol | 2 years
  Retrospective study based on recovering patient data from medical records

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France